CLINICAL TRIAL: NCT03844386
Title: A Phase I Pilot Study to Evaluate the Safety and Immunogenicity of the HIV-1 Vaccines MVA.tHIVconsv3 (M3) and MVA.tHIVconsv4 (M4) Given Alone or In Combination in HIV-1-Infected Adults Suppressed on Antiretroviral Therapy - The M&M Study
Brief Title: Study to Assess Safety and Ability to Induce Immune Responses of HIV-1 Vaccines M3 and M4 Given Alone or in Combination in HIV-infected Adults
Acronym: M&M
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-2502; U01AI131310-01 (NIH); IGHID 11810 (Other: University of North Carolina at Chapel Hill)
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Results first posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-07

CONDITIONS: HIV-1 Infection
Keywords: HIV-1; Infection; Suppressed; ART; Vaccines; Alone; Combination; Immunogenicity
MeSH Terms: conditions — Infections | interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 7(M3):7(M4):7(M3+M4):3(Placebo) to one of four study arms, and receive study treatment or placebo at Day 0.
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study in which both the participant and the investigator are blinded to what the participant receives.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MVA.tHIVconsv3 (M3) (Experimental): Participants in this arm receive one vaccine dose of MVA.tHIVconsv3 (M3) given IM at Day 0
  Interventions: Biological: MVA.tHIVconsv3
- MVA.tHIVconsv4 (M4) (Experimental): Participants in this arm receive one vaccine dose of MVA.tHIVconsv4 (M4) given IM at Day 0
  Interventions: Biological: MVA.tHIVconsv4
- MVA.tHIVconsv3 (M3)+MVA.tHIVconsv4 (M4) (Experimental): Participants in this arm receive a single combined dose containing each vaccine type MVA.tHIVconsv4 (M3) + MVA.tHIVconsv4 (M4) given IM at Day 0
  Interventions: Biological: MVA.tHIVconsv3; Biological: MVA.tHIVconsv4
- Placebo (Placebo Comparator): Participants in this arm receive one saline (placebo) dose given IM at Day 0
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MVA.tHIVconsv3 — viral-vector, MVA, expressing immunogens derived from conserved yet immunogenic regions of HIV-1
  Other Names: M3
  Arms: MVA.tHIVconsv3 (M3); MVA.tHIVconsv3 (M3)+MVA.tHIVconsv4 (M4)
Biological: MVA.tHIVconsv4 — viral-vector, MVA, expressing immunogens derived from conserved yet immunogenic regions of HIV-1
  Other Names: M4
  Arms: MVA.tHIVconsv3 (M3)+MVA.tHIVconsv4 (M4); MVA.tHIVconsv4 (M4)
Other: Placebo — The appropriate amount of Sodium Chloride for Injection USP, 0.9% will be drawn into a syringe.
  Other Names: Normal saline, Sodium Chloride
  Arms: Placebo

SUMMARY:
This is a double blind, randomized, placebo-controlled, parallel design, study in which 24 HIV-infected participants with durable viral suppression will be randomly assigned to receive vaccination with MVA.tHIVconsv3 (M3), MVA.tHIVconsv4 (M4), M3+M4 combined, or placebo. Participants will be randomized 7:7:7:3 to one of four study arms, and receive study treatment or placebo at Day 0. Each enrolled participant will complete the study in approximately 33.5 weeks (8.4 months).

The purpose of this study is to find out:

* If it is safe for people to receive injections of two investigational HIV vaccines, called MVAtHIVconsv3 and MVAtHIVconsv4 alone or in combination.
* If giving participants these vaccine doses will increase their immune system's ability to kill HIV virus.

DETAILED DESCRIPTION:
This is a Phase 1, single site, pilot study to evaluate the safety and immunogenicity of the M3 and M4 vaccines administered alone or in combination in HIV-infected participants suppressed on ART.

This is a double blind, randomized, placebo-controlled, parallel design study to evaluate the safety and immunogenicity of viral-vector, MVA, expressing immunogens, tHIVconsv3 (M3) and tHIVconsv4 (M4), derived from conserved yet immunogenic regions of HIV-1. The participant population is HIV-1 infected adults suppressed on ART with plasma HIV-1 RNA <50 copies/mL.

Hypotheses: The administration of M3 or M4 or M3+M4 together will be safe in HIV-1-infected participants suppressed on ART. The simultaneous administration of M3 with M4 (M3+M4) will result in both an increase in total magnitude of HIV-1-specific T cell responses and increase the breadth of T cells targeting conserved regions of HIV-1 compared with either M3 or M4 vaccination alone.

The vaccine and placebo doses will be administered to all participants as an IM (intramuscular) injection in the deltoid muscle of the non-dominant arm, unless a participant requests vaccination in their dominant arm. Participants continue their baseline ART regimen throughout the study. Randomized assignment 7:7:7:3 occurs at Day 0 to one of four arms as provided below:

Arm 1 - 7 participants - Treatment: M3 - Dose (pfu): 2x10-8 - Route: IM; Arm 2 - 7 participants - Treatment: M4 - Dose (pfu): 2x10-8 - Route: IM; Arm 3 - 7 participants - Treatment: M3+M4 - Dose (pfu): 1x10-8, each vaccine - Route: IM; Arm 4 - 3 participants - Treatment: Placebo/saline - Dose: N/A - Route: IM; M3 = MVA.tHIVconsv3; M4 = MVA.tHIVconsv4; pfu = plaque forming units; IM = intramuscular

The primary safety outcome is the occurrence of at least one ≥ Grade 3 Adverse Event (AE) including signs/symptoms, lab toxicities, and/or clinical events that are possibly, probably, or definitely related to study treatment through 28 days following vaccination. The primary safety analysis will be blinded through Day 28 after the last dose of vaccine/placebo and the second leukapheresis is completed by the last participant.

Screening, Enrollment, and Leukapheresis. The participant reviews and signs the informed consent (ICF). Participants meeting eligibility requirements enroll and undergo one leukapheresis procedure between Day -60 and Day 0. The leukapheresis procedure collects white blood cells allowing for completion of detailed immunologic and virologic assays with minimal blood loss. Participants have the option to consent to a lymph node FNA; participants choosing this option will complete the pre-vaccine FNA between Day -60 and Day 0 and a post-vaccine FNA between Day 7 and Day 21. The post-vaccine FNA should be collected even if the pre-vaccine collection attempt is unsuccessful.

Randomization, Study Treatment, Follow-up Assessment, and Leukapheresis. Randomization occurs at Day 0 when a randomization identification number (RID) will be assigned. All participants receive a vaccine or placebo dose as an IM injection. Post vaccination safety assessments occur via clinical evaluations, and lab testing/evaluations. The study will collect research assays at designated visits.

At Day 28, all participants will undergo their 2nd leukapheresis. This procedure can be completed between Day 21 through Day 35. The leukapheresis product will be used for immunologic and virologic research assays post vaccine/placebo. Participants will be followed for immunogenicity assessments through Day 70 and safety assessments through Day 168 (Week 24) following the administration of vaccine/placebo at Day 0.

Note: The post-vaccine leukapheresis must be done as close to Day 28 as possible. There may be a rare situation where the completion of the procedure in the 2-week visit window will not be possible. As soon as the study coordinator becomes aware of this scenario, the study coordinator should notify the study PI (or designee) to schedule the procedure outside the study window, preferably earlier (between Days 14 and 28). If the procedure can only be done after Day 35, participants should complete the Day 28 visit with collection of a 42.5 mL ACD sample at that visit.

ELIGIBILITY:
Inclusion Criteria:

1. HIV infection documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral assay.

   A reactive initial rapid test should be confirmed by either another type of rapid assay or an E/CIA that is based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a Western blot or a plasma HIV-1 RNA viral load.

   WHO (World Health Organization) and CDC (Centers for Disease Control and Prevention) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment.
2. Ages ≥ 18 to ≤ 65 years old
3. Able and willing to give written informed consent.
4. Able and willing to provide adequate locator information.
5. Able and willing to comply with time requirements for protocol-specified visits and evaluations.
6. Able and willing to commit to all study visits including follow-up through Day 168 (Week 24).
7. Continuous ART prior to screening, defined as not missing more than 9 total days and never more than 4 consecutive days in the last 3 months.
8. On a stable ART regimen defined as no changes in any ART medication within the 30 days prior to screening.
9. Permitted ART regimens include:

   * 1) At least 3 ART agents (not counting ritonavir or cobicistat as one of the agents if less than a 200mg total daily dose). One of the agents must include an integrase inhibitor, NNRTI (Non-Nucleoside Reverse Transcriptase Inhibitors), or a boosted-PI (protease inhibitor).

   OR
   * 2) Two ART agents in which one of the agents is either a boosted protease inhibitor or an integrase inhibitor.

   NOTE: Other potent fully suppressive antiretroviral combinations will be considered on a case-by-case basis.

   NOTE: Changes in drug formulation or dose are allowed (e g, TDF to TAF, ritonavir to cobicistat or separate ART agent dosing to fixed-dose combination), but none within 30 days prior to screening.

   NOTE: Prior changes in, or elimination of, medications for easier dosing schedule, intolerance, toxicity, an improved side effect profile or within a drug class are permitted if an alternative suppressive regimen was maintained, but not within 30 days prior to screening.
10. Ability and willingness of participant to continue ART throughout the study.
11. Plasma HIV-1 RNA <50 copies/mL at 3 time points in the previous 24 months prior to screening and never ≥50 copies/mL on 2 consecutive time points in the last 24 months.
12. At least 1 documented HIV-1 RNA result <50 copies/mL ≥24 months but ≤ 36 months prior to screening.
13. Plasma HIV-1 RNA level <50 copies/mL on an FDA-approved HIV RNA assay performed at a US CLIA Certified Laboratory (or its equivalent) at screening.
14. CD4 cell count ≥ 350 cells/mm3, performed at any US laboratory that has a CLIA certification or its equivalent at screening.
15. Hepatitis C (HCV) antibody negative result at screening or, if the participant is HCV antibody positive, a negative HCV RNA at screening.
16. Hepatitis B surface antigen (HBsAg) negative at screening.
17. Adequate vascular access for leukapheresis.
18. Able and willing to receive IM injections without difficulty.
19. All women must have a negative serum pregnancy test at screening regardless of reproductive potential.

    Note: The serum pregnancy test must have a sensitivity of at least 25 mIU/mL.
20. All participants must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization, egg donation) while on study and for 4 months after their vaccination.

    Note: Women of child bearing potential is defined as women who have not been post-menopausal for at least 24 consecutive months, i.e., who have had menses within the preceding 24 months, or women who have not undergone surgical sterilization, specifically hysterectomy and/or bilateral oophorectomy or bilateral salpingectomy
21. All men and women participating in sexual activity that could lead to pregnancy must agree to consistently use at least one of the following forms of birth control for at least 21 days prior to Visit 4 (Day 0) and for 4 months after their vaccination:

    * Condoms (male or female) with or without a spermicidal agent
    * Diaphragm or cervical cap with spermicide
    * Intrauterine device (IUD)
    * Tubal ligation
    * Hormone-based contraceptive

    NOTE: For female participants receiving ritonavir or cobicistat, estrogen-based contraceptives are not reliable and an alternative method should be suggested.
22. Men and women who are not of reproductive potential are eligible without requiring the use of contraceptives. Acceptable documentation detailing sterilization and menopause are specified below.

    Note: Men who have sex with men only will not be required to use contraception.

    Written or oral documentation communicated by clinician or clinician's staff of one of the following:
    * Physician report/letter
    * Operative report or other source documentation in the patient record (a laboratory report of azoospermia is required to document successful vasectomy)
    * Discharge summary
    * Follicle stimulating hormone-release factor (FSH) measurement elevated into the menopausal range as established by the reporting laboratory
23. Agrees not to enroll on another study of an investigational research agent during the study period.

    NOTE: Investigational research agent is defined as any unlicensed investigational drug not yet approved for use in humans.
24. Willingness to defer routine vaccination except for influenza and COVID-19 from within the previous 28 days of screening through 28 days after vaccination at Day 0.

    NOTE: Potential participants should delay enrollment on study until 14 days after receiving the influenza and/or COVID-19 vaccine.
25. Adequate organ function as indicated by the following laboratory values:

Hematological: Absolute neutrophil count (ANC) ≥ 1,000 /mcL; Platelets ≥ 100,000/mcL; Hemoglobin ≥ 12 g/dL (male) and ≥ 11.5 g/dL (females)

Coagulation: Prothrombin Time or INR<1.1 x ULN (upper limit of normal)

Chemistries: Serum potassium levels within normal limits; Serum magnesium levels1; Glucose - Screening serum glucose ≤ Grade 1 (fasting or non-fasting)

1 = LLN for Mg++ per the clinical laboratory's normal range used for this study is a grade 1 event per the DAIDS Toxicity Table and is allowed for eligibility.

Renal: Creatinine clearance determined by the CKD-Epi equation - eGFR > 60mL/min

Hepatic: Serum total bilirubin - Total bilirubin <1.1 x ULN. If total bilirubin is elevated, direct bilirubin must be <2 x ULN

If the participant is on an atazanavir -containing therapy then a direct bilirubin should be measured instead of the total bilirubin and must be ≤1.0mg/dL.

AST (SGOT) and ALT (SGPT)<1.25 X ULN Alkaline Phosphatase <1.25 X ULN

Urinalysis: Protein < 2+; Blood < 2+ (for women, before or after menses) LLN = lower limit of normal; UPN = upper limit of normal; WNL = within limit of normal

Exclusion Criteria:

1. If the HIV provider or study investigator is unable, as assessed by the study PI or protocol team, to construct a fully active alternative regimen based on previous resistance testing and/or treatment history.
2. Women of childbearing age/potential must not be breast feeding, pregnant, or planning pregnancy any time from enrollment to 4 months after vaccination at Day 0.
3. Body Mass Index (BMI) ≥40 kg/m2
4. Untreated syphilis infection (defined as a positive rapid plasma reagin (RPR) without clear documentation of treatment).

   NOTE: In cases of untreated syphilis, participant may rescreen following documentation of adequate treatment of syphilis.
5. Current treatment for HCV with antiviral therapy or participants who have received HCV treatment within 6 months prior to screening.
6. HIV RNA ≥150 copies/mL in the 6 months prior to screening.
7. Received any infusion blood product, immune globulin, or hematopoetic growth factors within 6 months prior to screening.
8. Use of any of the following within 90 days prior to screening: immunomodulatory, cytokine, or growth stimulating factors such as systemic cytotoxic chemotherapy, , immune globulin, interferon, cyclosporine, methotrexate, azathioprine, anti-CD25 antibody, IFN, interleukins, interleukin-2 (IL-2), hydroxyurea, thalidomide, sargramostim (granulocyte macrophage-colony stimulating factor [GM-CSF]), growth factors, dinitrochlorobenzene (DNCB), thymosin alpha, thymopentin, inosiplex, polyribonucleoside, or diticarb sodium, coumadin, warfarin, or other Coumadin derivative anticoagulants.
9. Intent to use immunomodulators (e.g., IL-2, IL-12, interferons or TNF modifiers) during the course of the study.
10. Use of systemic corticosteroids or topical steroids over a total area exceeding 15 cm2 within 30 days prior to screening, or anticipated need for periodic use of corticosteroids during the study.

    NOTE: For participants receiving ritonavir or cobicistat, (either as a booster or protease inhibitor [PI]) as part of their ART regimen, the concomitant use of oral/systemic/topical/inhaled/ intranasal corticosteroids is prohibited.
11. Use of any prior HIV vaccine (prophylactic and/or therapeutic) or HIV immunotherapy.

    Note: exceptions allowed for antibody therapies per PI review and approval.

    Note: exceptions allowed for IGHID 11627 (UNC IRB 17-0468; NCT 03212989) per PI review and approval provided there is greater than 12 months since receipt of study-provided treatment.
12. Any experimental non-HIV vaccination within 1 year prior to screening.

    NOTE: the receipt of an FDA Emergency Use Authorization (EUA) sanctioned COVID-19 vaccine is not considered exclusionary and should be reviewed with the protocol PI on a case-by-case basis.
13. Prior immunization with a recombinant Adenovirus or MVA vaccine

    Note: Prior immunization with smallpox vaccine is not exclusionary.

    NOTE: This exclusion INCLUDES COVID-19 vaccines with adenovirus vector (i.e., Janssen and AstraZeneca).
14. Live attenuated vaccines received within 60 days prior to screening (i.e., varicella; measles, mumps, rubella [MMR]; yellow fever, oral polio, shingles).

    NOTE: Individuals who require vaccination will delay screening for the study until 60 days after receiving the injection.
15. History of prior IgG therapy or immunization with any experimental immunogens (antibodies) within 6 months of screening.
16. Use of any investigational treatment within 6 months prior to screening, with the exception of Phase II studies of antiretroviral agents.

    NOTE: Co-enrollment with other studies under an IND using an FDA approved medication that are not otherwise listed as prohibited will be considered on a case-by-case basis.

    NOTE: The receipt of an FDA Emergency Use Authorization (EUA) sanctioned COVID-19 vaccine or treatment will be reviewed with the protocol PI and will be considered on a case-by-case basis.
17. For any serious illness requiring systemic treatment or hospitalization, the participant must either complete therapy or be clinically stable on therapy, in the opinion of the site investigator, for at least 90 days prior to screening.
18. Treatment for an active HIV-related opportunistic infection within 90 days prior to screening.
19. History of malignancy within the last 5 years.

    NOTE: A history of non-melanoma skin cancer (e.g., basal cell carcinoma or squamous cell skin cancer) is not exclusionary with documentation of topical treatment or of complete resection at least 3 months prior to screening).
20. Immune deficiency other than that caused by HIV infection.
21. Any medical, psychiatric, occupational or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence or assessment of safety.
22. Hypertension - Exclude for blood pressure consistently > 150 mm Hg systolic and >100 mm Hg diastolic.

    Note: Elevated BP occurring during research leukapheresis procedures completed within the past 12 months are excluded from this requirement. Isolated elevations must be noted as acceptable and signed by study PI or designee.
23. History of auto-immune disease, including Type I diabetes mellitus, with specific exception of:

    * Vitiligo
    * Resolved childhood atopic dermatitis
    * Psoriasis (with the exception of psoriatic arthritis) not requiring systemic treatment (within the past 2 years).
    * Grave's disease with subsequent return to a euthyroid state (clinically and by laboratory testing).
24. Seizure disorder: History of seizure(w) within the past 3 years. Also exclude if participant has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
25. History of unexplained syncope or fainting episodes within 12 months of study screening.
26. History of Asplenia - absence of normal spleen function as indicated by:

    * Splenectomy
    * Sickle cell disease
27. Bleeding disorder including factor deficiency, coagulopathy or platelet disorder that requires special precautions (easy bruising without a formal diagnosis is not exclusionary).
28. Allergy to eggs and/or egg products.
29. History of anaphylaxis or severe adverse reaction to vaccines including symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain.
30. History of hereditary angioedema, acquired angioedema or idiopathic angioedema.
31. Known or suspected hypersensitivity to any vaccine component.
32. Unstable asthma (e.g. sudden acute attacks occurring without an obvious trigger) or asthma requiring:

    * Daily steroid or long acting beta-agonist prevention
    * Hospitalization in the last two years
33. Depo-provera injection at the site of administration (upper left or right medial deltoid muscles) within the 3 months prior to screening, if other deltoid is not an option.
34. History of allergy to latex.
35. Active chronic skin problems such as eczema or psoriasis.
36. Known psychiatric or substance abuse disorder/dependence that, in the opinion of the site investigator, would interfere with cooperation with the requirements of the trial.
37. Compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric illness or a physical illness, e.g., infectious disease.
38. Prisoner recruitment and participation is not permitted.
39. Inability to communicate effectively with study personnel.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2022-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L Gay, MD, MPH, Principal Investigator — UNC-Chapel Hill; Nilu Goonetilleke, PhD, Principal Investigator — UNC-Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants in this arm receive one saline (placebo) dose given IM at Day 0
  Placebo: The appropriate amount of Sodium Chloride for Injection USP, 0.9%
Period: Overall Study
Arm/Group | MVA.tHIVconsv3 (M3) | MVA.tHIVconsv4 (M4) | MVA.tHIVconsv3 (M3)+MVA.tHIVconsv4 (M4) | Placebo
Started | 7 | 7 | 8 | 4
Completed Day 28 | 7 | 7 | 8 | 3
Completed | 7 | 7 | 7 | 3
Not Completed | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MVA.tHIVconsv3 (M3) | MVA.tHIVconsv4 (M4) | MVA.tHIVconsv3 (M3)+MVA.tHIVconsv4 (M4) | Placebo | Total
Number analyzed (Participants) | 7 | 7 | 8 | 4 | 26
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 43 [33 to 57] | 46 [31 to 58] | 36 [29.5 to 50] | 29.5 [26 to 41.5] | 41 [30 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 0 | 3
  Male | 5 | 6 | 8 | 4 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 3
  Not Hispanic or Latino | 6 | 6 | 7 | 4 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 6 | 1 | 14
  White | 3 | 3 | 2 | 3 | 11
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 7 | 8 | 4 | 26
Baseline CD4 Cell Count [Median (Full Range); unit: cells/mm^3] | 690 [534 to 1169] | 679 [412 to 1379] | 804.5 [442 to 1431] | 740 [562 to 1157] | 742.5 [412 to 1431]
Baseline HIV-1 RNA PCR Level [Median (Full Range); unit: copies/ml] | 30 [20 to 100] | 20 [20 to 40] | 40 [20 to 40] | 40 [20 to 40] | 40 [20 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With a Grade 3 or Higher Treatment-Related Adverse Event (AE)
Description: The DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017 will be used to measure safety where Grade 3 is defined as severe and Grade 4 is defined as potentially life-threatening. Treatment-Related AEs will be assessments that are considered related to study product as possible, probable, or definite as defined in the protocol.
Time Frame: First day of study treatment through 28 days following vaccination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MVA.tHIVconsv3 (M3) | MVA.tHIVconsv4 (M4) | MVA.tHIVconsv3 (M3)+MVA.tHIVconsv4 (M4) | Placebo
Number analyzed (Participants) | 7 | 7 | 8 | 4
percentage of participants | 43 [10 to 81] | 14 [0 to 58] | 0 [0 to 64] | 0 [0 to 60]

2. Secondary Outcome: Percent of Participants With a Grade 1 or Higher Treatment-Related Adverse Event (AE)
Description: The DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017 will be used to measure safety where Grade 1 is defined as mild, Grade 2 is defined as moderate, Grade 3 is defined as severe, and Grade 4 is defined as potentially life-threatening. Treatment-Related AEs will be assessments that are considered related to study product as possible, probable, or definite as defined in the protocol.
Time Frame: First day of study treatment through Day 168 (Week 24) following vaccination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MVA.tHIVconsv3 (M3) | MVA.tHIVconsv4 (M4) | MVA.tHIVconsv3 (M3)+MVA.tHIVconsv4 (M4) | Placebo
Number analyzed (Participants) | 7 | 7 | 8 | 4
percentage of participants | 100 [59 to 100] | 100 [59 to 100] | 100 [63 to 100] | 75 [19 to 99]

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent throughout treatment, a total of approximately 24 weeks.
Arm/Group | MVA.tHIVconsv3 (M3) | MVA.tHIVconsv4 (M4) | MVA.tHIVconsv3 (M3)+MVA.tHIVconsv4 (M4) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7 | 8/8 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MVA.tHIVconsv3 (M3) (N=7) | MVA.tHIVconsv4 (M4) (N=7) | MVA.tHIVconsv3 (M3)+MVA.tHIVconsv4 (M4) (N=8) | Placebo (N=4)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 4 (4) | 4 (4) | 3 (3) | 0 (0)
Fatigue (General disorders) | 4 (7) | 5 (5) | 5 (5) | 2 (2)
Influenza like illness (General disorders) | 4 (7) | 2 (2) | 4 (4) | 1 (1)
Injection site discoloration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 6 (13) | 6 (12) | 8 (13) | 2 (3)
Injection site swelling (General disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Malaise (General disorders) | 5 (9) | 5 (5) | 3 (3) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tissue infiltration (General disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Vessel puncture site hemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Citrate toxicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Post procedural contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural hypertension (Injury, poisoning and procedural complications) | 6 (12) | 7 (13) | 7 (15) | 4 (5)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood HIV RNA increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 3 (3) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 5 (7) | 4 (4) | 1 (1)
Dizziness (Nervous system disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 6 (9) | 4 (4) | 5 (5) | 3 (3)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT03844386/Prot_SAP_000.pdf